CLINICAL TRIAL: NCT03964870
Title: Spanish Registry of RYR1 and CACNA1S Polymorphisms in Unselected Population for Evaluation of Malignant Hyperthermia Susceptibility (MHS). RYCA Registration
Brief Title: Spanish Registry of RYR1 and CACNA1S Polymorphisms
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Principal Investigator of Anesthesiology, Hospital Universitario La Fe
Other Study IDs: RYCA
Record Dates: First submitted 2019-05-22; First posted 2019-05-28 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Malignant Hyperthermia; Polymorphisms in Genes RYR1 and CACNAS1S
Keywords: Malignant Hyperthermia
MeSH Terms: conditions — Malignant Hyperthermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples to identify genes RYR1 and CACNAS1S
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Diagnostic of polymorphisms in malignant hyperthermia — Identify and catalogue the variants or polymorphisms in the RYR1 and CACNA1S genes in the Spanish population.

SUMMARY:
Study design: The Spanish registry of RYR1 and CACNA1S polymorphisms (RYCA) is an anonymous descriptive observational multicentre study that aims to identify and catalogue the variants or polymorphisms in the RYR1 and CACNA1S genes in the Spanish population. Secondarily, its correlation with the binding mutations described in both genes at European level by the EMHG will be evaluated to assess the incidence of malignant hyperthermia in Spain. The RYCA registry complies with the highest standards of European and international homologation, both with regard to computer security and the protection of personal data (Data Protection Law 15/1999).

Hypothesis: Performing a Spanish registry of RYR1 and CACNA1S polymorphisms will contribute to describe the variants present in our environment and determine their relationship with MH susceptibility.

Objectives:

* Describe the national polymorphisms of the RYR1 and CACNA1S genes
* To evaluate the incidence of genetic MH susceptibility according to the recommendations of the EMHG.

The presence of polymorphisms in a population that has not been studied before may have a difficult correlation with the mutations described in the EMHG webpage.

Eligibility Criteria: The sample contained in the registry will originate from the genetic data of patients unrelated to HM who have been sequenced the RYR1 and CACNA1S gene by another pathology. The data related to the genetic analysis will be provided without identifying data of the patient or the clinical history. There will be no possibility of identification of the patient by the team responsible for the RYCA registry, so the request for informed consent is not viable. There will be no selection of participants or patient follow-up.

Methodology: A preliminary pilot study will be conducted in an unselected anonymous cohort of the sequenced exome database of the RYR1 and CACNA1S gene at the La Fe Health Research Institute (IISlaFe). The population contained in this database is random and unrelated to HM and the patients are anonymous, so we do not have access to personal data or medical history. If the analysis is feasible, a request for collaboration will be transferred to the Genetics Services / Research Units with experience in the exome sequencing of the RYR1 and CACNA1S genes. Anonymous readings will be requested to carry out the registration and description of the variants existing in the Spanish population and their relationship with the variants described by the EMHG.

Variables: The registry will include the chromosomal coordinates, number of total patients included, number of patients whose variant is in heterozygosis, number of patients whose variant is in homozygosis and allelic frequency. Thus, for each of the genes of interest, and making use of their respective chromosomal coordinates, information regarding the variants that these might include will be extracted.

Sample size. Sample size calculation is not considered since it is a descriptive record.

ELIGIBILITY:
The sample contained in the registry will originate from the genetic data of patients unrelated to malignant hyperthermia who have been sequenced the RYR1 and CACNA1S gene by another pathology. The data related to the genetic analysis will be provided without identifying data of the patient or the clinical history. There will be no possibility of identification of the patient by the team responsible for the RYCA registry, so the request for informed consent is not viable. There will be no selection of participants or patient follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria: Patents with malignant hyperthermia which genes RYR1 and CACNA1S have been sequenced for another pathology
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-11-05 (Estimated); Study Completion 2020-12-05 (Estimated)

PRIMARY OUTCOMES:
Describe the national polymorphisms of the RYR1 and CACNA1S genes | Day 1
  The peripheral blood must be extracted by venous puncture. For this, it is necessary to carry out the extraction of the blood by qualified health personnel respecting the corresponding hygienic-sanitary norms. The blood must be in a tube with EDTA anticoagulant (preferably). The method of extraction of peripheral blood DNA: is carried out mainly by automatic procedure using the QIASYMPHONY SP DNA extractor-purifying equipment and the QYASIM DNA MIDI KIT Kit (Qiagen), Cat. No: 931255, following the manufacturer's protocols.
  The DNA extraction stage is collected in the GESTLAB system as SAMPLE PROCESSING (it comprises extraction and quantification via Nanodrop, as indicated below).
To evaluate the incidence of genetic MH susceptibility according to the recommendations of the EMHG. | Day 1
  The peripheral blood must be extracted by venous puncture. For this, it is necessary to carry out the extraction of the blood by qualified health personnel respecting the corresponding hygienic-sanitary norms. The blood must be in a tube with EDTA anticoagulant (preferably). The method of extraction of peripheral blood DNA: is carried out mainly by automatic procedure using the QIASYMPHONY SP DNA extractor-purifying equipment and the QYASIM DNA MIDI KIT Kit (Qiagen), Cat. No: 931255, following the manufacturer's protocols.
  The DNA extraction stage is collected in the GESTLAB system as SAMPLE PROCESSING (it comprises extraction and quantification via Nanodrop, as indicated below).

CONTACTS AND LOCATIONS:
Locations (1):
- IIS la Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No